CLINICAL TRIAL: NCT02446184
Title: Fetal Cystoscopy for Severe Lower Urinary Tract Obstruction - a Prospective Trial
Brief Title: Fetal Cystoscopy for Lower Urinary Tract Obstruction
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Original P.I. of this study transferred to a different institution.
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Michael Belfort, MD PhD, Professor Baylor College of Medicine and Co-Director Texas Children's Fetal Center, Baylor College of Medicine
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BCM H33626
Record Dates: First submitted 2015-05-12; First posted 2015-05-18 (Estimated); Last update posted 2017-02-13 (Actual); Status verified 2017-02

CONDITIONS: Urethral Obstruction
Keywords: urethral obstruction; posterior urethral valves; lower urinary tract obstruction
MeSH Terms: conditions — Urethral Obstruction

STUDY DESIGN:
Intervention Model Description: This study is an un-blinded, non-randomized, single arm Phase 1 study. Fetal intervention is usually offered to patients carrying fetuses with isolated LUTO that meet the inclusion criteria. Once the patient elected to have fetal intervention, fetal cystoscopy will be offered as an experimental procedure as an option to fetal vesico-amniotic shunting.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Fetal cystoscopy (Experimental): Fetal cystoscopy will be performed under maternal local anesthesia and fetal anesthesia. The dilated posterior urethra will be directly evaluated. Laser fulguration will be performed in case of posterior urethral valves. However, if a non membrane-like structure is found, even with the fluid injection or the guide-wire, urethral atresia (UA, US or Prune Belly syndrome) will be diagnosed and we will not attempt to perforate this structure. A vesicoamniotic shunting placement will be performed in this situation depending on the patient's consent prior to the surgery.
  Interventions: Procedure: Fetal Cystoscopy
- Vesicoamniotic shunt (Active Comparator): The fetal vesicoamniotic shunt is considered the standard prenatal therapy for severe LUTO. Amnioinfusion and vesicoamniotic shunt placement will be performed under ultrasound guidance.
  Interventions: Procedure: Fetal vesicoamniotic shunt
- No fetal intervention group (No Intervention): Those patients that refuse fetal intervention and do not elect to terminate the pregnancy will be followed as part of the no fetal intervention group.

INTERVENTIONS:
Procedure: Fetal Cystoscopy — Fetal cystoscopy will be performed under maternal local anesthesia and fetal anesthesia. The dilated posterior urethra will be directly evaluated. Laser fulguration will be performed in case of posterior urethral valves. However, if a non membrane-like structure is found, even with the fluid injection or the guide-wire, urethral atresia (UA, US or Prune Belly syndrome) will be diagnosed and we will not attempt to perforate this structure. A vesicoamniotic shunting placement will be performed in this situation depending on the patient's consent prior to the surgery.
  Arms: Fetal cystoscopy
Procedure: Fetal vesicoamniotic shunt — Fetal vesicoamniotic shunt will be performed under ultrasound guidance
  Other Names: Bladder shunt
  Arms: Vesicoamniotic shunt

SUMMARY:
This is a pilot study to evaluate the safety, feasibility, and effectiveness of fetal cystoscopy as an experimental procedure in avoiding perinatal death and renal impairment and to compare to the investigators clinical experience with fetal vesicoamniotic shunting.

DETAILED DESCRIPTION:
Patients with severe LUTO will come for clinical evaluation as part of the standard clinical care at the Fetal Center at Texas Children's Hospital. Once the diagnosis of fetal severe LUTO is confirmed and the patient is considered for fetal intervention, patient will be invited to participate in the present study. Fetal cystoscopy will be offered as an optional experimental procedure.

The following information will be obtained in the standard clinical care visit as usual: a. demographics (maternal age, parity); b. gestational age at the diagnosis of LUTO; c. fetal ultrasound findings including documentation of cervical length, gestational age,fetal bladder size, bladder wall thickness, degree of fetal hydronephrosis, amount of amniotic fluid, fetal biometry; d. fetal urinary biochemistry; e. fetal echocardiogram findings.

The standard management options for fetal LUTO include expectant management, fetal vesico-amniotic shunting or termination of pregnancy according to the law. These options will be offered to all patients as the first set of management options and the gold standard. In addition, the investigators group will offer the procedure as an alternative experimental option, with a full explanation of the experimental nature of the procedure, the technical benefits and difficulties, and the risks and potential benefits of the procedure and the limited long-term outcomes information. Those patients who request participation in the present study will be informed that they can, a priori, select a crossover arm if for any reason the fetal cystoscopic procedure is not possible. They can elect that a fetal vesico-amniotic shunting be performed or prenatal expectant management or even termination of pregnancy (as part of the standard management of fetuses with LUTO).

Participation in the study:

Once the patient is deemed eligible, all prenatal standard management options will be offered first to the patient. Fetal cystoscopy will be offered as an investigational procedure for evaluation. If the patient opts for the fetal cystoscopy, we will explain that this procedure can be diagnostic and therapeutic. In order to prevent coercion, the investigation procedure will be presented to the patient in a manner that is an option and voluntary, if the patient chooses not to participate in the investigational procedure, the clinical care will not be affected. Informed consent to participate in the present study will be obtained. We will also include non-English speaking subjects in the present study. We will submit a full Spanish consent via amendment for IRB approval after approval of the English consent. We will not enroll any non-English subjects until we receive final approval. The study flow is demonstrated in Figure 1 (see attached document).

Description of the fetal cystoscopy procedure (experimental procedure):

Fetal cystoscopy will be performed between 16 0/7 and 25 6/7 weeks at the Pavilion for Women - TCH. This procedure will be performed under maternal local anesthesia and sedation. In some cases, according to the anesthesiologist's indication, maternal epidural may be performed. Fetal anesthesia will be performed by ultrasound-guided injection into fetal arm or leg of a combination of fentanyl (15µglKg), atropine and vecuronium (0.5-2mg/Kg).

Prophylactic tocolysis will be used in all patients with a protocol employing magnesium sulfate - 6 gram IV loading dose followed by a 2 gram/hour continuous infusion for 24 hours, followed by nifedipine 10mg Q6 during until 36 weeks of gestation.

Prophylactic antibiotics will also be used during the procedure using Cefazolin 2 g IV immediately before the procedure. Nafcillin will be injected into the amniotic cavity at the conclusion of the procedure. In case the patient has allergies to cephalosporin, clindamycin 600 mg will be used as alternative.

Steroids for fetal lung maturation will be given between 24 and 25 6/7 weeks (two doses of 12 mg betamethasone given 24 hours apart, with the last dose given 48-72 hours before the procedure), if the procedure is performed during this gestational period.

The procedure will be performed percutaneously under ultrasound-fetoscopic guidance. An 18G needle will be introduced into the fetal bladder through the maternal abdominal wall and uterus under ultrasound guidance. Using a Seldinger technique an 8-9Fr Cook trocar will be inserted through the maternal wall towards the fetal bladder. A curved Storz sheath for 1.3 mm (11530AA, Karl Storz, Tuttlinglen, Germany) or 2.0 mm fetoscopy (26120BA, Karl Storz, Tuttlingen, Germany) or flexible ureteroscope will be introduced into the Cook catheter into the fetal bladder. After confirming that the trochar is inside the fetal bladder, urine samples will be collected for further renal function analysis. The fetoscope will be advanced toward the bladder neck and the dilated posterior urethra. If a membrane-like obstruction of the urethral lumen is seen, the diagnosis of PUV will be confirmed and at this time the valves will be fulgurated using a Diode laser with low energy (15-20W). If necessary, we will use a guide-wire to perforate the valves. Fulguration of the valves will be performed very cautiously with the laser fiber almost touching them in order to avoid damaging peripheral tissues. When the valves are completely disrupted, the urine will be released through the now patent urethra, which results in emptying the bladder. A transurethral shunt may be placed depending on the cause of the obstruction (urethral stenosis). In addition, power Doppler will be applied to confirm passage of fluid through the patent urethra into the amniotic cavity. However, if a non membrane-like structure is found, even with the fluid injection or the guide-wire, urethral atresia (UA, US or Prune Belly syndrome) will be diagnosed and we will not attempt to perforate this structure. A vesicoamniotic shunting placement will be performed in this situation depending on the patient's consent prior to the surgery.

The postsurgical care is going to follow the same standard prenatal care after fetal vesico-amniotic shunting. The expected hospital course is 72 hours as it is also expected for fetal vesico-amniotic shunting; however, it is possible that the patient will be hospitalized for complications or preterm labor. The patient will then be discharged home with recommendations for modified bed rest for the first 2 weeks post discharge, but will subsequently be allowed to graduate to moderate activity if the uterus is quiescent. Patients will return on a weekly basis for clinical and ultrasound evaluation. On ultrasound, fetal kidneys, bladder thickness and dilatation, and amniotic fluid volume will be assessed. Fetal Surveillance by biophysical profiles and Doppler studies will begin at 34 weeks

Delivery mode will be performed based on the obstetrical management following the investigators clinical algorithm.

The subjects that undergo fetal cystoscopy will have exactly the same postnatal routine (standard of care) clinical follow-up that is provided to all infants with LUTO. All infants with LUTO are followed-up by the pediatric urology and nephrology services and may need postnatal surgical intervention. At birth, the clinical evaluation will include a renal ultrasound, voiding cysto-urethrogram (VCUG) as well as clinical laboratory examinations such as serum creatinine, sodium, calcium, potassium and chloride, and a urine analysis will be performed as part of the standard clinical care. Information from these routine examinations will be collected and documented.

ELIGIBILITY:
Inclusion Criteria:

* Fetus with LUTO, dilated bladder, "keyhole sign" and bilateral hydronephrosis
* Oligohydramnios or Anhydramnios after 18 weeks
* "Favorable urine analysis after 18 weeks (urinary sodium is < 100mEq/L, chloride < 90mEq/L, osmolarity <200mOsm/L and β2-microglobulin <6mg/L 7)
* Absence of chromosomal abnormalities and associated anomalies (Normal karyotype by invasive testing (amniocentesis or CVS))
* Gestational age at the time of the procedure will be between 16 0/7 weeks and 25 6/7 weeks

Exclusion Criteria:

* Fetal anomaly unrelated to LUTO
* Congenital cardiac anomaly
* Increased risk for preterm labor including short cervical length (<1.5 cm), history of incompetent cervix with or without cerclage, and previous preterm birth
* Placental abnormalities (previa, abruption, accreta) known at time of enrollment - A body-mass index ≥ 35
* Contraindications to surgery including previous hysterotomy in active uterine segment
* Technical limitations precluding fetoscopic surgery, such as uterine fibroids, fetal membrane separation, uterine anomalies incompatible with fetoscopy
* Maternal-fetal Rh isoimmunization, Kell sensitization or neonatal alloimmune thrombocytopenia affecting the current pregnancy
* Maternal HIV, Hepatitis-B, Hepatitis-C status positive because of the increased risk of transmission to the fetus during maternal-fetal surgery. If the patient's HIV or Hepatitis status is unknown, the patient must be tested and found to have negative results before enrollment
* Maternal medical condition that is a contraindication to surgery or anesthesia
* Patient does not have a support person (ie. Spouse, partner, mother) available to support the patient for the duration of the pregnancy at Texas Children's Hospital/Ronald McDonald House
* Patient does not have healthy insurance to cover routine clinical care at Texas Children's Hospital including prenatal care, prenatal ultrasound, amniocentesis, tocolysis, admission, delivery, and fetal vesico-amniotic shunting. The exception will be fetal cystoscopy which is considered an experimental procedure.
* Inability to comply with the travel and follow-up requirements of the trial
* Participation in another intervention study that influences maternal and fetal morbidity and mortality or participation in this trial in a previous pregnancy
* Patients declining invasive testing
* Family does not meet psychosocial criteria.

Ages: 16 Weeks to 26 Weeks | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 8 (Actual)
Dates: Start 2014-12-04 (Actual); Primary Completion 2016-08 (Actual); Study Completion 2016-08-23 (Actual)

PRIMARY OUTCOMES:
Postnatal survival at 2 years of life | 2 years
  We will evaluate the survival rate at 2 years of life

SECONDARY OUTCOMES:
Postnatal renal function at 2 years of life | 2 years
  We will evaluate the renal function at 2 years of life based on the glomerular filtration rate (GFR). In addition, we will evaluate the need for dialysis and renal transplant.

CONTACTS AND LOCATIONS:
Overall Officials: Michael A Belfort, MD, PhD, Principal Investigator — Baylor College of Medicine; Rodrigo Ruano, MD, PhD, Principal Investigator — Baylor Colleg of Medicine (Previously); Mayo Clinic (currently)
Locations (1):
- Texas Children's Hospital Pavilion for Women, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ruano R, Pimenta EJ, Duarte S, Zugaib M. Four-dimensional ultrasonographic imaging of fetal lower urinary tract obstruction and guidance of percutaneous cystoscopy. Ultrasound Obstet Gynecol. 2009 Feb;33(2):250-2. doi: 10.1002/uog.6292. No abstract available. PMID 19173237
- [Result] Ruano R, Duarte S, Bunduki V, Giron AM, Srougi M, Zugaib M. Fetal cystoscopy for severe lower urinary tract obstruction--initial experience of a single center. Prenat Diagn. 2010 Jan;30(1):30-9. doi: 10.1002/pd.2418. PMID 19967749
- [Result] Ruano R, Yoshisaki CT, Salustiano EM, Giron AM, Srougi M, Zugaib M. Early fetal cystoscopy for first-trimester severe megacystis. Ultrasound Obstet Gynecol. 2011 Jun;37(6):696-701. doi: 10.1002/uog.8963. PMID 21337440
- [Result] Morris RK, Ruano R, Kilby MD. Effectiveness of fetal cystoscopy as a diagnostic and therapeutic intervention for lower urinary tract obstruction: a systematic review. Ultrasound Obstet Gynecol. 2011 Jun;37(6):629-37. doi: 10.1002/uog.8981. Epub 2011 May 16. PMID 21374748
- [Result] Ruano R. Fetal surgery for severe lower urinary tract obstruction. Prenat Diagn. 2011 Jul;31(7):667-74. doi: 10.1002/pd.2736. Epub 2011 Mar 17. PMID 21413041
- [Result] Ethun CG, Zamora IJ, Roth DR, Kale A, Cisek L, Belfort MA, Haeri S, Ruano R, Welty SE, Cassady CI, Olutoye OO, Cass DL. Outcomes of fetuses with lower urinary tract obstruction treated with vesicoamniotic shunt: a single-institution experience. J Pediatr Surg. 2013 May;48(5):956-62. doi: 10.1016/j.jpedsurg.2013.02.011. PMID 23701767
- [Result] Ruano R, Yoshizaki CT, Giron AM, Srougi M, Zugaib M. Cystoscopic placement of transurethral stent in a fetus with urethral stenosis. Ultrasound Obstet Gynecol. 2014 Aug;44(2):238-40. doi: 10.1002/uog.13293. Epub 2014 Jun 26. PMID 24375864
- [Result] Sananes N, Favre R, Koh CJ, Zaloszyc A, Braun MC, Roth DR, Moog R, Becmeur F, Belfort MA, Ruano R. Urological fistulas after fetal cystoscopic laser ablation of posterior urethral valves: surgical technical aspects. Ultrasound Obstet Gynecol. 2015 Feb;45(2):183-9. doi: 10.1002/uog.13405. PMID 24817027
- [Result] Ruano R, Sananes N, Sangi-Haghpeykar H, Hernandez-Ruano S, Moog R, Becmeur F, Zaloszyc A, Giron AM, Morin B, Favre R. Fetal intervention for severe lower urinary tract obstruction: a multicenter case-control study comparing fetal cystoscopy with vesicoamniotic shunting. Ultrasound Obstet Gynecol. 2015 Apr;45(4):452-8. doi: 10.1002/uog.14652. Epub 2015 Mar 2. PMID 25157756